CLINICAL TRIAL: NCT03102112
Title: Noninvasively Predicting Isocitrate Dehydrogenase Gene Status in Glioma by Amide Proton Transfer Imaging
Brief Title: Noninvasively Predicting Gene Status of Glioma
Acronym: NPGSOG
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDLL-20151013
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Glioma of Brain
Keywords: Glioma APT MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with glioma: Consecutive patients with privious MRI scans or symptoms that suggested a cerebral mass, not yet receive treatment.
  Interventions: Other: MRI examination

INTERVENTIONS:
Other: MRI examination — A noninvasive medical diagnostic technique in which the absorption and transmission of high-frequency radio waves are analysed as they irradiate the hydrogen atoms in water molecules and other tissue components placed in a strong magnetic field. This computerized analysis provides a powerful aid to the diagnosis and treatment planning of many diseases, including cancer.

SUMMARY:
Malignant gliomas are the most common and deadly primary brain tumors in adults. The clinical outcome of patients with glioblastoma depends on key molecular genetic alteration. Specifically, Isocitrate Dehydrogenase Gene Mutation, an independent favorable prognostic factor, serve as diagnostic and prognostic markers of glioma. Thus, accurate grading of a glioma is fundamental in order to determine the treatment strategy. Amide proton transfer (APT) imaging is a noninvasive molecular MRI technique based on chemical exchange saturation transfer mechanism that detects endogenous mobile proteins and peptides in biological tissues. Preliminary studies have shown that APT-weighted (APTw) signal intensity could serve as a new imaging biomarker, by revealing significantly higher signal intensities in the high-grade gliomas compared with the low-grade gliomas. The purpose of this study was to investigate the value of amide proton transfer imaging (APT) in the noninvasive evaluation of isocitrate dehydrogenase (IDH) gene status in glioma.

DETAILED DESCRIPTION:
Materials and Methods:

The whole brain MRI examinations were performed on a 3.0-T MRI system (Discovery MR750, General Electric Medical System, Milwaukee, WI, USA) with an eight-channel head coil (General Electric Medical System). Conventional MRI, contrast-enhanced MRI, DWI and amide proton transferimaging were performed in regular sequence during the same examination. Finally, contrast-enhanced T1-weighted spin echo sequence was acquired in the transverse, sagittal, and coronal planes after intravenous administration of 0.01 mmol/kg gadodiamide (Omniscan; GE Healthcare, Co. Cork, Ireland).

MRI data processing and image analysis:

All data were transferred to a workstation (Advantage Workstation 4.6, General Electric Medical System, Milwaukee, Wisconsin, USA) for processing.The MR imaging of all the patients were assessed independently by two experienced neuroradiologist (HYC and YLF, who have 12 and 6 years of experience, respectively, in neurologic-oncologic imaging) who were blinded to the patient's information. Next, a region of interest (ROI) was drawn manually on the solid part of the tumor with the relatively higher signal intensity on APT image.

Statistical analysis:

Categorical data obtained from image were calculated using the Fisher's exact test. Quantitative data were denoted as the mean and standard deviation. The Kolmogorov-Smirnov (K-S) test was used to assess the normality of data distribution.APT-weighted (APTw) signal intensity were tested for differences between the IDH mutation and the IDH wild-type by using independent sample t test.

ELIGIBILITY:
Inclusion Criteria:

* no hypertension or cerebral vascular diseases
* no use of corticosteroid drugs
* no MRI contraindication
* no allergic constitution

Exclusion Criteria:

* pregnant wowan
* motion cause poor image quality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients and out patients with head MRI scans and symptoms that suggested a cerebral mass.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-10 (Estimated); Study Completion 2018-03-03 (Estimated)

PRIMARY OUTCOMES:
APT image for assessing the gene alteration | 15 months
  Prospectively acquire the APTw signal intensity to assess the efficiency for predicting the ATRX as prognostic or predictive biomarkers of gliomasloss/mutation, 1p/19q status, IDH1/2 gene mutations and MGMT promoter methylation

SECONDARY OUTCOMES:
APT image for predicting the survival of glioma | 24 months
  to find the correlation coefficient between the APTw signal intensity and the survival of patients with glioma

CONTACTS AND LOCATIONS:
Overall Officials: Yu Han, MD, Principal Investigator — Department of Radiology, Tangdu Hospital, the Fourth Military Medical University
Locations (1):
- Yu han, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided